CLINICAL TRIAL: NCT05815992
Title: Accuracy of the Characterization of Adnexal Masses, Indeterminate at Ultrasonography, Using a Magnetic Resonance Imaging Protocol Without Contrast: Validation of the Cambridge Score
Brief Title: Accuracy of the Characterization of Adnexal Masses, Indeterminate at Ultrasonography, Using a MRI Protocol Without Contrast: Validation of the Cambridge Score
Acronym: CAMBRIDGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4298
Record Dates: First submitted 2023-03-29; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Adnexal Mass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective observational study is to evaluate the accuracy and to validate the Cambridge Score,a Test Index to predict the malignancy of the ovarian lesions on the basis of an MRI examination without contrast

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Indeterminate adnexal masses at the ultrasonography;
* Signed Informed Consent.

Exclusion Criteria:

* Diagnosis of an extraovary mass;
* Synchronous tumors;
* Previous history of neoplasy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with indeterminate adnexal masses can be included.
Study Population: Patients with a diagnosis of indeterminate adnexal masses after ultrasonography that will undergo to an MRI examination can be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of generalizability of the Cambridge Score through external validations | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Evaluation of Cambridge Score when diagnosed by different readers | Through study completion, an average of 3 years
Evaluation of diagnostic agreement between the Non-contrast and contrast-enhanced MRI | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy